CLINICAL TRIAL: NCT03770169
Title: Validation of Patient Reported Outcome Measures for Use in Vulvodynia
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: D-FR-52120-252
Record Dates: First submitted 2018-11-29; First posted 2018-12-10 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of this project is to demonstrate content validity and usability of the modified Vulvar Pain Assessment Questionnaire (mVPAQ), the modified Female Sexual Function Index (mFSFI), and pain on intercourse Numeric Rating Scale (NRS) for adult patients with Vulvodynia

ELIGIBILITY:
Inclusion Criteria:

* Fluent in understanding, speaking and reading US-English
* Have vulvodynia with pain for at least 6 months

Exclusion Criteria:

* Clinically significant history of alcohol/drug abuse or dependence within the last 2 years

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects referred by clinicians
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Validation of mVPAQ | 1 week
  Cognitive debrief and usability through interviews and completion of an electronic diary
Validation of mFSFI | 1 week
  Cognitive debrief and usability through interviews and completion of an electronic diary
Validation of Pain on Intercourse Numeric Rating Scale (NRS) | 1 week
  Cognitive debrief and usability through interviews and completion of an electronic diary. Pain on Intercourse NRS that describes pain experienced during this sexual intercourse episode by number. The higher is the number the worse is pain.

SECONDARY OUTCOMES:
Vulvar pain NRS | 1 week
  Assess understanding of the appropriateness of the vulvar pain NRS through interview and completion of an electronic diary

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (4):
- United States (4):
  - San Diego Sexual Medicine, San Diego, California
  - Center for Vulvovaginal Disorders, Washington D.C., District of Columbia
  - Omaha OB-GYN Associates, PC, Omaha, Nebraska
  - The Center for Vulvovaginal Disorders, New York, New York